CLINICAL TRIAL: NCT06499935
Title: The Immediate Effects of Rigid Taping Versus Kinesio-Taping on Plantar Pressure Distribution in Basketball Players With Chronic Ankle Instability
Brief Title: The Effect of Taping on Plantar Pressure Distribution in Players With Chronic Ankle Instability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed ElMelhat, Associate Professor of Physical Therapy, Cairo University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Taping on Foot Pressure
Record Dates: First submitted 2024-06-29; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Ankle Injuries; Ankle Injuries and Disorders; Ankle Sprains
MeSH Terms: conditions — Ankle Injuries; Disease

STUDY DESIGN:
Intervention Model Description: Phase 1:Observational study. Phase 2: Double-blinded randomized control trial study. An explanation of the procedure and a written consent form will be provided. Then the CAIT will be used followed by assigning the participants into a healthy group and an injured group for the observational part and collecting the data on the injured foot. Then further randomly divided the injured group into a rigid taping group, a sham taping group, and a control group. Application of the interventions will be done to the affected foot and sham tape will be applied to the control group then the effects will be observed and the measurements will be noted and compared to the previous data. The CAIT will be used again to observe the differences that may result. The study will take place at Mousawat Institution.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rigid Taping Group (Experimental): A single application of tape will be fastened to the fibula's lateral malleolus, extended beneath the foot, and crossed the medial foot at the calcaneus and navicular tuberosity. After that, it will wrapped around the fibular and tibial shafts and passed across the anterior part of the ankle. The tape will be applied similarly to the other application, with 1.5 inches of overlap between the strips.
  Interventions: Other: Rigid Taping
- Kinesio Taping Group (Experimental): Elastic kinesiology tape will be employed in this investigation. Patients will be comfortably positioned on a table raised sufficiently so that their feet couldn't contact the ground. At the hindfoot, a 2-inch, 25-centimeter strip will be applied, stretching it seventy-five percent from the middle third of the medial tibia to the fibula (lateral malleolus), around the calcaneus. Applying the strip in the maximally supinated position while going in the direction mentioned will allow the foot to eventually reach its maximum dorsal flexion. The interior aspect of the tibial bone and fibula will then wrapped
  Interventions: Other: Kinesio-Taping
- Sham Taping Group (Sham Comparator): There are two steps to Sham taping: The internal malleolus is the starting point of the first stage, which extends to the lower limb's inner middle point. The second stage starts at the external malleolus and extends to the lower limb's outer middle point.
  Interventions: Other: Sham Taping

INTERVENTIONS:
Other: Rigid Taping — It is usually light brown or beige and is designed to hold firm, making it ideal for providing support or stability to a joint.
  Arms: Rigid Taping Group
Other: Kinesio-Taping — Kinesio Taping Method is a therapeutic tool utilised by rehabilitation specialists in all programs. Kinesio Taping Method utilises four types of Kinesio Tex Tapes, each with specific properties designed for use on fragile, sensitive skin or applied with higher tensions.
  Arms: Kinesio Taping Group
Other: Sham Taping — Sham taping is the use of any type of tape in a random and ineffective fashion for the purposes of comparison with other taping techniques and types.
  Arms: Sham Taping Group

SUMMARY:
The goal of this study is to investigate whether there exists a difference in baropdometric readings of plantar pressure between individuals with chronic ankle instability and normal health individuals, in addition another goal of this study is to investigate the effect of rigid taping vs. kinesio taping on plantar pressure distribution as well as stability markers in individuals with chronic ankle instability.

The main questions aimed to answer are:

1. Is there a difference in plantar pressure distribution between individuals with chronic ankle instability and individuals without chronic ankle instability?
2. What effect do rigid and kinesio taping have on plantar pressure distribution and ankle stability markers?
3. Which tape affects plantar pressure distribution and ankle stability better?

Participants will:

Firstly be divided into two macro groups, one with chronic ankle instability and one without, with an observational part of the study to be carried out to investigate the differences in plantar pressure between both groups.

Secondly, the group with chronic ankle instability will be divided into two micro groups one receiving rigid taping and the other receiving kinesio taping, and the immediate effects of these tapes in terms of plantar pressure and ankle stability will be recorded and compared before and after within groups, and after between both groups.

DETAILED DESCRIPTION:
Basketball players frequently suffer from lateral ankle sprains and multiple repetitions can cause chronic ankle instability. The authors contend that professional basketball can no longer be regarded as a noncontact sport because of the rising rate of injuries to players in the league. An orthopedic strapping treatment for the foot called rigid taping involves applying tape along the plantar part of the foot and inferior to the malleoli.

Another type of taping method gives the musculoskeletal system external support, kinesio-taping has long been employed in the rehabilitation and prevention of sports-related injuries in athletes and sports participants. The goal of an anti-pronation taping technique is to constrain an overpronated foot by offering temporary external support.

Thus the aim of this study is to determine the immediate effects of rigid taping versus kinesio-taping on static and dynamic plantar pressure distribution in basketball players with chronic ankle instability. An explanation of the procedure and a written consent form will be provided, and the assessment will be taken at the beginning of the spring semester of 2024/2025 for inclusion and exclusion. Then the CAIT will be used followed by assigning the participants into a healthy group and an injured group for the observational part and collecting the data on the injured foot. Then further randomly divided the injured group into AP, LD, and a control group. Application of the interventions will be done to the affected foot and sham tape will be applied to the control group then the effects will be observed and the measurements will be noted and compared to the previous data. The CAIT will be used again to observe the differences that may result. The study will take place at Mousawat Institution.

ELIGIBILITY:
Inclusion Criteria:

* A history of at least 1 significant ankle sprain
* The initial sprain must have occurred at least 12 months before study enrollment
* A history of the previously injured ankle joint "giving way" and/or recurrent sprain and/or "feelings of instability."
* Cumberland Ankle Instability Tool: score of 24 or less

Exclusion Criteria:

* A history of previous surgeries to the musculoskeletal structures (i.e., bones, joint structures, nerves) in either lower extremity
* A history of a fracture in either lower extremity requiring realignment
* Acute injury to musculoskeletal structures of other joints of the lower extremity in the previous 3 months that impacted joint integrity and function (i.e., sprains, fracture) resulting in at least 1 interrupted day of desired physical activity.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2024-09-25 (Estimated); Study Completion 2024-10-25 (Estimated)

PRIMARY OUTCOMES:
Baropodometric measurements of plantar pressure distribution. | immediately after the intervention
  The plantar pressure data will be measured during single-leg stance and natural walk using the Gaitview (®) AFA-50 system (alFOOTs, Seoul, Republic of Korea). The pressure platform included a 410 × 410 × 3 mm active area consisting of a 45-mm thick floor mat (700 × 500 mm), comprising 2,304 (48 × 48) force-sensitive resistor sensors and sampling data at 17 Hz (Kim et al., 2012). An investigation of the reliability of the Gaitview® system using the two-step gait-initiation method was done. It demonstrated good to moderate reliability for measuring plantar pressure, and that it is suitable for use in clinical and research trials (Kim et al., 2012). Data will be recorded and saved using the same device.

SECONDARY OUTCOMES:
Ankle Stability | immediately after the intervention
  Cumberland ankle instability Tool (CAIT) will be completed for each participant to measure the functional ankle instability severity. The CAIT consists of 9 items each containing choices ranging from 1 to 6, with scores from 0 to 5 for the right foot and left foot separately where the maximum score is 30 indicating high functional ankle stability while the minimum score is 0 indicating severe functional ankle instability (Hiller et al., 2006).

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed M. El Melhat, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided